CLINICAL TRIAL: NCT03070327
Title: A Phase I Trial of B-cell Maturation Antigen (BCMA) Targeted EGFRt/BCMA-41BBz Chimeric Antigen Receptor (CAR) Modified T Cells With or Without Lenalidomide for the Treatment of Multiple Myeloma (MM)
Brief Title: BCMA Targeted CAR T Cells With or Without Lenalidomide for the Treatment of Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-025
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
Keywords: B-cell Maturation Antigen (BCMA); Targeted EGFRt/BCMA-41BBz; Chimeric antigen receptor (CAR); Lenalidomide; 17-025
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; Lenalidomide

STUDY DESIGN:
Intervention Model Description: This is an open-label, dose escalating, nonrandomized, single-center, phase I study of EGFRt/BCMA-41BBz CAR T cells in patients with a diagnosis of MM. Dose escalation will follow a standard 3-by-3 escalation design. Cohorts of 3-6 patients will be infused with escalating doses of EGFRt/BCMA-41BBz CAR T cells to establish the maximum tolerated dose (MTD). After a dose level has been determined safe to escalate (DLT in 0/3 or 1/6 patients), a parallel cohort at that dose level will be conducted while patients are taking Lenalidomide.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BCMA Targeted CAR T Cells with or without Lenalidomide (Experimental)
  Interventions: Biological: EGFRt/BCMA-41BBz CAR T cell; Drug: Cyclophosphamide; Drug: Lenalidomide.

INTERVENTIONS:
Biological: EGFRt/BCMA-41BBz CAR T cell — Modified T cell infusions will be administered 2-7 days following the completion of conditioning chemotherapy.There are 3 planned dose levels for this study: 1x10^6, 3x10^6, and 1x10^7 EGFRt/BCMA-41BBz CAR T cells/kg, and a dose -1 level at 3x10^5 EGFRt/BCMA-41BBz CAR T cells/kg, if needed; each dose cohort will consist of 3-6 patients.
Drug: Cyclophosphamide — Cyclophosphamide 3000 mg/m2 IV once on day -7 to -2 or low intensity cy/flu (cyclophosphamide 300 mg/m2/day x 3 + fludarabine 30 mg/m2/day x 3) with the last day occurring on day -7 to -2 are the default options for is the default conditioning chemotherapy.
Drug: Lenalidomide. — A cohort of patients will be treated with CAR T cell therapy and concomitant Lenalidomide. 10mg PO 21/28 days will be started no less then 1 week prior to clinical apheresis.

SUMMARY:
The purpose of this phase I clinical trial is to test the safety of these CAR T cells in patients with myeloma.

There are two parts of this study. Part 1 of the study consists of screening for BCMA, Lenalidomide assignment and cell collection. Part 2 of the study is treatment with modified CAR T cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed MM by MSKCC pathologist, with MM cells expressing BCMA, previously treated with 2+ prior lines of therapy including an IMiD and a PI, either with refractory, persistent, or progressive disease
* Age ≥ 18 years of age
* Creatinine ≤2.0 mg/dL, direct bilirubin ≤2.0 mg/dL, AST and ALT ≤3.0x upper limit of normal (ULN)
* Adequate pulmonary function as assessed by ≥92% oxygen saturation on room air by pulse oximetry.
* HGB≥7g/dl, ANC≥1,000/mm3, Platelet≥30,000/mm3 without transfusion or growth factor support for at least 1 week
* M spike ≥0.5 g/dL or involved free light chain ≥10 mg/dL with an abnormal free light chain ratio

Exclusion Criteria:

* Karnofsky performance status <70
* Pregnant or lactating women. Women and men of childbearing age should use effective contraception while on this study and continue for 1 year after all treatment is finished
* Impaired cardiac function (LVEF <40%) as assessed by ECHO or MUGA scan
* Patients with following cardiac conditions will be excluded:

  * New York Heart Association (NYHA) stage III or IV congestive heart failure
  * Myocardial infarction ≤6 months prior to enrollment
  * History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
  * History of severe non-ischemic cardiomyopathy
* Patients with HIV or active hepatitis B or hepatitis C infection are ineligible
* Patients with any concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation or hormonal therapy, with the exception of squamous and basal cell carcinoma of skin
* Patients with a prior allogeneic transplant ARE eligible UNLESS previously or currently experienced GvHD that required systemic steroids or other systemic lymphotoxic therapy
* Patients on systemic steroids (except if solely for adrenal replacement) within two weeks of collection
* Active auto-immune disease including connective tissue disease, uveitis, sarcoidosis, inflammatory bowel disease, or multiple sclerosis, or have a history of severe (as judged by the principal investigator) autoimmune disease requiring prolonged immunosuppressive therapy
* Prior treatment with gene modified T cells
* Prior or active CNS involvement by myeloma (eg leptomeningial disease). Screening for this, for example, by lumbar puncture, is only required if suspicious symptoms or radiographic findings are present
* Plasma cell leukemia
* Pre-existing (active or severe) neurologic disorders (e.g. pre-existing seizure disorder)
* Active uncontrolled acute infections
* Any other issue which, in the opinion of the treating physician, would make the patient ineligible for the study
* Patients who previously had any intolerance to Lenalidomide 10 mg or who have a contraindication to Lenalidomide will not be eligibile for concominant treatment with Lenalidomide but will remain eligible for CAR T cell therapy without Lenalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
MTD of gene-modified T cells | 36 months
  The MTD is defined as the highest dose with an observed incidence of DLT in no more than one out of six patients treated at a particular dose level. T cell dose may be divided in up to three infusions administered over up to 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Sham Mailankody, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Jain T, Knezevic A, Pennisi M, Chen Y, Ruiz JD, Purdon TJ, Devlin SM, Smith M, Shah GL, Halton E, Diamonte C, Scordo M, Sauter CS, Mead E, Santomasso BD, Palomba ML, Batlevi CW, Maloy MA, Giralt S, Smith E, Brentjens R, Park JH, Perales MA, Mailankody S. Hematopoietic recovery in patients receiving chimeric antigen receptor T-cell therapy for hematologic malignancies. Blood Adv. 2020 Aug 11;4(15):3776-3787. doi: 10.1182/bloodadvances.2020002509. PMID 32780846
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm